CLINICAL TRIAL: NCT06610266
Title: Efficacy and Safety of Weifuchun Tablet in Reversing Gastric Intestinal Metaplasia: A Multi-center, Open-label, Randomized Controlled Trial
Brief Title: Efficacy and Safety of Weifuchun Tablet in Reversing Gastric Intestinal Metaplasia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yongquan Shi (Other)
Responsible Party: Sponsor-Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20242224-F-1
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Gastric Intestinal Metaplasia
MeSH Terms: interventions — weifuchun; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Weifuchun tablet group (Experimental): Patients in the Weifuchun tablet group will receive oral Weifuchun tablet at a dosage of 1400 mg three times daily for 6 months.
  Interventions: Drug: Weifuchun
- The folic acid group (Active Comparator): Patients in the folic acid group will receive oral folic acid at a dosage of 5 mg three times daily for 6 months.
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: Weifuchun — Subjects will be instructed to take four tablets (1400mg) of Weifuchun three times daily, and visit the hospital every 4 weeks for evaluation of the subjective symptoms and to receive a new supply of medication.
  Arms: The Weifuchun tablet group
Drug: Folic Acid — Subjects will be instructed to take one tablet (5mg) of folic acid three times daily, and visit the hospital every 4 weeks for evaluation of the subjective symptoms and to receive a new supply of medication.
  Arms: The folic acid group

SUMMARY:
The goal of this clinical trial is to investigate the efficacy and safety of Weifuchun tablet in treating gastric intestinal metaplasia in Helicobacter pylori-negative adults. The main questions it aims to answer are: Does Weifuchun tablet promote the regression of gastric intestinal metaplasia in individuals without Helicobacter pylori infection? What medical problems do participants experience when taking Weifuchun tablet? Researchers will compare the effectiveness of Weifuchun tablet in treating gastric intestinal metaplasia with that of folic acid, as suggested by the Chinese consensus on management of gastric epithelial precancerous conditions and lesions (2020). Participants will: Take Weifuchun tablets or folic acid every day for 6 months. Visit the clinic once every 4 weeks for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 18 to 75 years old.
* patients with OLGIM stage Ⅱ-Ⅳ diagnosed by upper gastrointestinal endoscopy and histopathological examination within the last 3 months.
* patients without Helicobacter pylori infection, including patients who had successful Helicobacter pylori eradication before enrollment.

Exclusion Criteria:

* a history of regular use (defined as at least once per week) of non-steroidal anti-inflammatory drugs (NSAIDs) and/or statins.
* a history of stomach surgery (including endoscopic submucosal dissection and endoscopic mucosal resection) or previously diagnosed malignant tumor.
* a history of heart failure, renal failure, liver cirrhosis or chronic hepatic failure; patients with contraindications or allergies to the drugs in this study.
* breastfeeding or pregnancy.
* a history of substance abuse or alcohol abuse within the past one year.
* patients with severe mental illness.
* refusal to undergo drug treatment.
* refusal to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The regression rate of gastric intestinal metaplasia based on OLGIM stage in different groups. | From enrollment to the end of treatment at 6 months.
  Regression was defined as a OLGIM stage decreased at least one grade.
The progression rate of gastric intestinal metaplasia based on OLGIM stage in different groups. | From enrollment to the end of treatment at 6 months.
  Progression was defined as a OLGIM stage increased at least one grade.

SECONDARY OUTCOMES:
The regression rate of gastric atrophy based on OLGA stage in different groups. | From enrollment to the end of treatment at 6 months.
  Regression was defined as a OLGA stage decreased at least one grade.
The progression rate of gastric atrophy based on OLGA stage in different groups. | From enrollment to the end of treatment at 6 months.
  Progression was defined as a OLGA stage increased at least one grade.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, China

IPD SHARING:
Plan to Share IPD: No